CLINICAL TRIAL: NCT03783013
Title: The Influence of Tomato Soy Juice on Inflammation in Overweight and Obese Adults
Brief Title: Tomato Juice for Health Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was halted prematurely because of research restrictions related to COVID-19
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS61 - Tomato Juice Study
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Soy and Low Lycopene Juice (Other): Participants will consume two cans daily of a low lycopene tomato juice in addition to a diet low in lycopene and isoflavones.
  Interventions: Other: Low Lycopene Tomato Juice
- Soy and Lycopene Juice (Other): Participants will consume two cans daily of a high lycopene tomato juice with added soy germ extract in addition to a diet low in lycopene and isoflavones.
  Interventions: Other: High Lycopene Tomato Juice With Soy Germ Extract

INTERVENTIONS:
Other: High Lycopene Tomato Juice With Soy Germ Extract — Tomato juice made from high lycopene tomatoes with soy germ extract added
  Arms: Soy and Lycopene Juice
Other: Low Lycopene Tomato Juice — Tomato juice made from low lycopene tomatoes with no soy germ extract added
  Arms: No Soy and Low Lycopene Juice

SUMMARY:
The primary objective of this study is to determine if tomato-soy juice can reduce inflammation, which is linked to chronic disease

DETAILED DESCRIPTION:
The aim of this study is to improve understanding of how diet can ameliorate the state of chronic inflammation. Short term inflammation is an important part of the body's response to injury, but long term inflammation, as happens in the state of obesity, can result in a multitude of secondary problems, like cancer, diabetes, and cardiovascular disease. Using a novel tomato-soy juice, we aim to demonstrate the potential of tomato-soy juice for reducing inflammation in adults.

ELIGIBILITY:
Inclusion Criteria:

* Between 30 and 75 years old
* Voluntarily agree to participate and sign an informed consent document

Exclusion Criteria:

* Aged < 30 years or > 75 years
* Known allergy or intolerance to tomatoes or soy
* BMI < 30 or > 45 kg/m2
* Blood plasma glucose > 125 mg/dL
* Blood plasma/serum triglycerides > 250 mg/dL
* Blood plasma/serum cholesterol > 240 mg/dL
* Diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Previous bariatric or gastrointestinal surgery affecting absorption
* Suspected or known strictures, fistulas or physiological/mechanical gastrointestinal obstruction
* Presence of gastrointestinal or malabsorptive disorders (including Crohn's, ileus or ulcerative colitis, or diverticulitis), or nutrient malabsorption disease (such as celiac disease)
* Presence of autoimmune disease, metabolic disease, liver disorders, or kidney disorders
* Diagnosis or treatment of certain cancers in the past 3 years
* Use of tobacco products or marijuana
* Daily use of anti-inflammatory drugs
* Use of antibiotics over the previous 3 months
* Colonoscopy within a month of the study start date or during the study
* Use of a carotenoid or isoflavone-containing or metabolism-altering supplement for the last 1 month
* Use of certain medications (prescription or over-the-counter) that may interfere with the study objectives
* Unable or unwilling to give informed consent or communicate with study staff
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 | Day 15 of the study
  Interleukin 6 (IL6) is a blood cytokine and an indicator of inflammatory status. IL6 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 6 | Day 43 of the study
  Interleukin 6 (IL6) is a blood cytokine and an indicator of inflammatory status. IL6 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 6 | Day 71 of the study
  Interleukin 6 (IL6) is a blood cytokine and an indicator of inflammatory status. IL6 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 6 | Day 99 of the study
  Interleukin 6 (IL6) is a blood cytokine and an indicator of inflammatory status. IL6 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 8 | Day 15 of the study
  Interleukin 8 (IL8) is a blood cytokine and an indicator of inflammatory status. IL8 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 8 | Day 43 of the study
  Interleukin 8 (IL8) is a blood cytokine and an indicator of inflammatory status. IL8 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 8 | Day 71 of the study
  Interleukin 8 (IL8) is a blood cytokine and an indicator of inflammatory status. IL8 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interleukin 8 | Day 99 of the study
  Interleukin 8 (IL8) is a blood cytokine and an indicator of inflammatory status. IL8 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Tumor Necrosis Factor Alpha | Day 15 of the study
  Tumor Necrosis Factor Alpha (TNF-a) is a blood cytokine and an indicator of inflammatory status. TNF-a will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Tumor Necrosis Factor Alpha | Day 43 of the study
  Tumor Necrosis Factor Alpha (TNF-a) is a blood cytokine and an indicator of inflammatory status. TNF-a will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Tumor Necrosis Factor Alpha | Day 71 of the study
  Tumor Necrosis Factor Alpha (TNF-a) is a blood cytokine and an indicator of inflammatory status. TNF-a will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Tumor Necrosis Factor Alpha | Day 99 of the study
  Tumor Necrosis Factor Alpha (TNF-a) is a blood cytokine and an indicator of inflammatory status. TNF-a will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Monocyte chemoattractant protein-1 | Day 15 of the study
  Monocyte chemoattractant protein-1 (MCP-1) is a signalling molecule and is part of the inflammatory process. MCP-1 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Monocyte chemoattractant protein-1 | Day 43 of the study
  Monocyte chemoattractant protein-1 (MCP-1) is a signalling molecule and is part of the inflammatory process. MCP-1 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Monocyte chemoattractant protein-1 | Day 71 of the study
  Monocyte chemoattractant protein-1 (MCP-1) is a signalling molecule and is part of the inflammatory process. MCP-1 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Monocyte chemoattractant protein-1 | Day 99 of the study
  Monocyte chemoattractant protein-1 (MCP-1) is a signalling molecule and is part of the inflammatory process. MCP-1 will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interferon Gamma | Day 15 of the study
  Interferon gamma (INF-g) is a signalling molecule and is part of the inflammatory process. INF-g will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interferon Gamma | Day 43 of the study
  Interferon gamma (INF-g) is a signalling molecule and is part of the inflammatory process. INF-g will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interferon Gamma | Day 71 of the study
  Interferon gamma (INF-g) is a signalling molecule and is part of the inflammatory process. INF-g will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.
Interferon Gamma | Day 99 of the study
  Interferon gamma (INF-g) is a signalling molecule and is part of the inflammatory process. INF-g will be measured to determine how the treatment is affecting inflammatory status. Cytokines are measured in units of pg/mL.

SECONDARY OUTCOMES:
Flavonoids/Isoflavones will be measured | Days 1, 15, 43, 71, 99 of the study
  Blood and Urine will be analyzed for flavonoids/isoflavones and their metabolites in units of nanomolar
Carotenoids will be measured | Days 1, 15, 43, 71, 99 of the study
  Blood will be analyzed for carotenoids and metabolites in units of mmolar
Identification of metabolites that change in blood and urine by metabolomics | Days 1, 15, 43, 71, 99 of the study
  Metabolomics is the simultaneous measurement of the many thousand small molecule metabolites. Chromatography separates the metabolites, which are then ionized, then the detector detects the number of ion hits for each ion, which reflects the amount (number of ions) of a particular compound. If the detector detects more of an ion in blood or urine after one treatment vs. another, then the position on the chromatogram (units of time in minutes) and the ratio of the mass (atomic mass units) to charge (unitless) of the compound will be compared to the 75,000 entries in the METLIN metabolite library to identify what the compound is.
Cytokine production by peripheral blood mononuclear cells | Day 1, 15, 43, 71, 99 of the study
  Peripheral blood mononuclear cells produce inflammation molecules called cytokines when exposed to an irritant (called the stimulant in the assay). Peripheral blood mononuclear cells will be stimulated with an irritant and cytokine production will be measured in units of pg/ml.
Blood total cholesterol | Day 1, 15, 43, 71, 99 of the study
  Total cholesterol will be measured in blood. Units will be mmol/L.
Blood LDL cholesterol | Day 1, 15, 43, 71, 99 of the study
  LDL cholesterol will be measured in blood. Units will be mmol/L.
Blood HDL cholesterol | Day 1, 15, 43, 71, 99 of the study
  HDL cholesterol will be measured in blood. Units will be mmol/L.
Blood triglycerides | Day 1, 15, 43, 71, 99 of the study
  Triglycerides will be measured in blood. Units will be mmol/L.
Blood glucose | Day 1, 15, 43, 71, 99 of the study
  Glucose will be measured in blood. Units will be mmol/L.
Blood insulin | Day 1, 15, 43, 71, 99 of the study
  Insulin will be measured in blood. Units will be mmol/L.
Blood pressure | Day 1, 15, 43, 71, 99 of the study
  Blood pressure will be measured. Units will be mm Hg.
High Sensitivity c-Reactive Protein | Day 1, 15, 43, 71, 99 of the study
  High sensitivity c-reactive protein will be measured in blood. Units will be mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No